CLINICAL TRIAL: NCT02278588
Title: Effect of 2.5 Years of Rasagiline Therapy on Progression of Cognitive Biomarkers Assessed by MRI in Parkinson's Disease.
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Thomas Guttuso, Associate Professor of Neurology, Obstetrics & Gynecology, State University of New York at Buffalo
Other Study IDs: [616856-4]
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PD-R: Parkinson's disease receiving rasagiline
  Interventions: Drug: Rasagiline
- PD-NMAO: Parkinson's disease not receiving any MAO-B inhibitors
- HC: Healthy Controls

INTERVENTIONS:
Drug: Rasagiline
  Other Names: Azilect
  Groups: PD-R

SUMMARY:
In this investigator-initiated study, we will compare changes in brain cognitive biomarkers assessed by diffusion tensor imaging over 2.5 years among 12 patients with Idiopathic Parkinson's disease (IPD) receiving rasagiline, 20 IPD patients not receiving MAO-B inhibitors and 25 age-matched healthy controls. Will also compare the changes in Mini-Mental State Exam (MMSE) and Montreal Cognitive Assessment (MoCA) scores and plasma brain-derived neurotrophic factor (BDNF) with changes in brain cognitive biomarkers in all IPD patients and HC over 2.5 years.

ELIGIBILITY:
IPD or HC subjects who were enrolled in a similar study about 2.5 years ago and for whom Baseline DTI data are available.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Idiopathic Parkinson's disease (IPD) and Healthy Controls (HC)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in cognitive biomarkers assessed by DTI | 2.5 years
Comparison of change in cognitive biomarkers with change in MMSE and MoCA scores | 2.5 years

SECONDARY OUTCOMES:
Comparison of Baseline plasma BDNF with magnitude of change in brain cognitive biomarkers and MMSE and MoCA scores | 2.5 years
Comparison of changes in plasma BDNF with changes in brain cognitive biomarkers and MMSE and MoCA scores | 2.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States